CLINICAL TRIAL: NCT04230044
Title: A Post Marketing Observational Study to Evaluate the Safety and Efficacy of Fycompa® (Perampanel) as Add-on Therapy in Epilepsy Patients
Brief Title: A Study to Evaluate the Safety and Efficacy of Fycompa® (Perampanel) as Add-on Therapy in Participants With Epilepsy
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E2007-M065-411
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-11

CONDITIONS: Epilepsy; Partial-onset Seizures
Keywords: E2007; Fycompa; Perampanel; Partial onset seizures; Epilepsy; Seizures; Post marketing surveillance
MeSH Terms: conditions — Epilepsy; Seizures | interventions — perampanel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fycompa® (perampanel): Fycompa® (perampanel) (oral tablets) treatment will be initiated at 2 milligram (mg) once daily according to the approved package insert, as an add-on drug in addition to other anti-epileptic drugs (AEDs) as prescribed by physician. The dose will be increased based on clinical response and tolerability (by increments of 2 mg/day to a maintenance dose of 4 to 12 mg/day) and participants will be enrolled and observed prospectively for up to 54 Weeks.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — Perampanel tablets.
  Other Names: Fycompa; E2007

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of Fycompa® (perampanel) for the adjunctive treatment of partial-onset seizures with or without secondarily generalized seizures in participants with epilepsy aged 12 years and older.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged 12 years and older
2. Participants who were diagnosed with partial-onset seizures with or without secondarily generalized seizures.
3. Participants who were appropriate to receive Fycompa® as an adjunctive treatment participants starting at Visit 0 according to investigator's judgment.
4. Participants who had provided written informed consent

Exclusion Criteria:

1. Participants not fit to receive Fycompa® as per the latest prescribing information.
2. Participants who were participating in a clinical trial, at the time of the study.
3. Participants who showed evidence of clinically significant disease (cardiac, respiratory, gastrointestinal, renal disease, etc.) that in the opinion of the Investigators could affect the participant's safety or trial conduct.
4. Participants who according to the Investigators would not be able to comply with study procedures.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with epilepsy aged 12 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI) | Up to 54 Weeks
  AESI will include medication errors, lack of therapeutic efficacy, overdose, abuse, misuse, occupational exposure, paternal exposure and off label use, pregnancy, and exposure to drug during breast feeding.

SECONDARY OUTCOMES:
Change From Baseline in 28-day Seizure Count at the End of Treatment Period (Week 52) | Baseline, Week 52
Response Rate | Baseline, Week 12, Week 24 and Week 52
  Response rate will be defined as number of participants with response defined as more than or equal to (>=) 50 percent (%) reduction in 28-day seizure frequency from Baseline.
Change From Baseline in Clinical Global Impression of Change (CGIC) Scores | Baseline, Week 12, Week 24 and Week 52
  The CGIC is an assessment performed by the clinician, evaluating the change in the participant's symptoms over time. Assessment will be implemented based on frequency of seizure, severity of seizures, adverse events, and overall conditions on a 7-point scale with the scores as 1: very much improved, 2: much improved, 3: minimally improved, 4: no change, 5: minimally worse, 6: much worse, 7: very much worse.

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.